CLINICAL TRIAL: NCT00719602
Title: P1060 Substudy Comparing Differences in Malaria Parasitemia by Real Time Quantitative PCR in HIV-Infected Infants and Children on PI-Based HAART Versus NNRTI-Based HAART
Brief Title: Differences in Malaria Infection Levels in HIV-infected Infants and Children Receiving PI- and NNRTI-based HAART
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMPAACT P1068s; U01AI068632 (NIH)
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: HIV Infections; Malaria
Keywords: Coinfection
MeSH Terms: conditions — HIV Infections; Malaria; Coinfection | interventions — Lamivudine; Lopinavir; Nevirapine; Zidovudine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Previously received single-dose nevirapine (SD NVP); assigned to receive either an NNRTI- or PI-based regimen as a part of the study IMPAACT P1060
  Interventions: Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Nevirapine; Drug: Zidovudine
- 2 (Active Comparator): Have not previously received SD NVP; assigned to receive either an NNRTI- or PI-based regimen as a part of the study IMPAACT P1060
  Interventions: Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Nevirapine; Drug: Zidovudine

INTERVENTIONS:
Drug: Lamivudine — Taken orally twice daily
  Other Names: 3TC
Drug: Lopinavir/Ritonavir — Taken orally twice daily
  Other Names: LPV/r
Drug: Nevirapine — Taken orally twice daily
  Other Names: NVP
Drug: Zidovudine — Taken orally twice daily
  Other Names: ZDV

SUMMARY:
More than 1.5 million deaths of African children under 5 years of age have been due to Plasmodium falciparum malaria. When HIV and malaria are present as coinfections, they enhance each other's progression. The primary purpose of this study is to compare the malarial infection levels in HIV-infected infants and children receiving protease inhibitor (PI)- or non-nucleotide reverse transcriptase inhibitor (NNRTI)-based highly active antiretroviral therapy (HAART).

DETAILED DESCRIPTION:
The World Health Organization (WHO) reports 1 to 2 million malaria deaths annually, with most malaria-related deaths occurring in children. The malaria burden is compounded by the HIV epidemic, which is most prevalent in areas endemic for malaria, notably Sub-Saharan Africa where nine in ten children younger than 15 years of age are infected with HIV. The purpose of this study is to compare parasitemia levels in HIV-infected infants and children receiving PI- or NNRTI-based HAART regimens.

This study will enroll a total of 140 participants, 35 from each of the 4 groups in IMPAACT P1060.

This substudy will last until 24 weeks after the last P1060 enrollment or until P1060 study discontinuation. Participants must meet enrollment criteria for P1060 as well as additional criteria for this study. Study visits will occur as a part of P1060 study visits, all of which include a physical exam, blood collection, and assessments of HIV-related symptoms.

Participants are also encouraged to return to the primary clinic site for intercurrent illness visits for assessment, thick and thin blood smear, and filter paper blood collection, however these visits are not mandatory for study participation.

ELIGIBILITY:
Inclusion Criteria:

* Enrolling in study IMPAACT P1060
* Parent/legal guardian agrees to seek medical care for intercurrent illness at the study site, whenever possible, and agree to not use at-home remedies for febrile illness in the child

Exclusion Criteria:

None.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2009-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Parasitemia in blood samples | Throughout study

SECONDARY OUTCOMES:
Time of initiation of treatment for clinical malaria requiring conventional anti-malarial therapy | Throughout study
Severity of malarial disease | Throughout study
Measured anti-malaria IgG, protein in plasma, and mRNA transcripts in PBMC of chemokines | Throughout study
IL4-589C/T genotypes | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Hobbs, MD, Study Chair — NYU Langone Health; William Borkowsky, MD, Study Chair — NYU Langone Health
Locations (3):
- University of North Carolina Lilongwe (12001), Lilongwe, Malawi
- Makerere University - JHU Research Collaboration (30293), Kampala, Uganda
- George Clinic CRS (30273), Lusaka, Zambia

REFERENCES:
- [Background] Adetifa IM, Akinsulie AO, Temiye EO, Iroha EO, Ezeaka VC, Mafe AG, Grange AO. Effect of antiretroviral therapy on asymptomatic malaria parasitaemia in HIV-1 infected children. Niger Postgrad Med J. 2008 Jun;15(2):120-5. PMID 18575485
- [Background] Brahmbhatt H, Sullivan D, Kigozi G, Askin F, Wabwire-Mangenm F, Serwadda D, Sewankambo N, Wawer M, Gray R. Association of HIV and malaria with mother-to-child transmission, birth outcomes, and child mortality. J Acquir Immune Defic Syndr. 2008 Apr 1;47(4):472-6. doi: 10.1097/QAI.0b013e318162afe0. PMID 18332766
- [Derived] Hobbs CV, Gabriel EE, Kamthunzi P, Tegha G, Tauzie J, Petzold E, Barlow-Mosha L, Chi BH, Li Y, Ilmet T, Kirmse B, Neal J, Parikh S, Deygoo N, Jean Philippe P, Mofenson L, Prescott W, Chen J, Musoke P, Palumbo P, Duffy PE, Borkowsky W; P1068s Study Team. Malaria in HIV-Infected Children Receiving HIV Protease-Inhibitor- Compared with Non-Nucleoside Reverse Transcriptase Inhibitor-Based Antiretroviral Therapy, IMPAACT P1068s, Substudy to P1060. PLoS One. 2016 Dec 9;11(12):e0165140. doi: 10.1371/journal.pone.0165140. eCollection 2016. PMID 27936233